CLINICAL TRIAL: NCT01105923
Title: Making Accurate Problem Lists in the EHR
Brief Title: Study of an Intervention to Improve Problem List Accuracy and Use
Acronym: MAPLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Adam Wright, Senior Scientist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009P001846
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Asthma; COPD; Breast Cancer; Coronary Artery Disease; Congestive Heart Failure; Diabetes; Glaucoma; Hemophilia; Hypertension; Hyperthyroidism; Hypothyroidism; Myasthenia Gravis; Osteoporosis; Osteopenia; Renal Failure; Renal Insufficiency; Sickle Cell Disease; Stroke
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Asthma; Pulmonary Disease, Chronic Obstructive; Breast Neoplasms; Coronary Artery Disease; Heart Failure; Diabetes Mellitus; Glaucoma; Hemophilia A; Hypertension; Hyperthyroidism; Hypothyroidism; Myasthenia Gravis; Osteoporosis; Bone Diseases, Metabolic; Renal Insufficiency; Anemia, Sickle Cell; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receive CDS intervention (Experimental): Providers in clinics that will receive the CDS alert, as their clinic was randomized into our study.
  Interventions: Other: MAPLE
- No CDS intervention (No Intervention)

INTERVENTIONS:
Other: MAPLE — MAPLE is a CDS intervention within the EHR that will alert providers to problem lists gaps and present an opportunity to correct them.
  Arms: Receive CDS intervention

SUMMARY:
The aim of this study is to identify patients with problem list gaps and intervene to correct these gaps by creating clinical decision support interventions that alert providers to likely problem list gaps and offer clinicians the opportunity to correct them. The investigators will randomize the clinics that will receive the intervention and formally evaluate the study after a period of 6 months for improved problem list completeness to determine the effectiveness of our intervention.

DETAILED DESCRIPTION:
The clinical problem list is a cornerstone of the problem-oriented medical record. Problem lists are used in a variety of ways throughout the process of clinical care. In addition to its use by clinicians, the problem list is also critical for decision support and quality measurement.

Patients with gaps in their problem list face significant risks. For example, if a hypothetical patient has diabetes properly documented, his clinician would receive appropriate alerts and reminders to guide care. Additionally, the patient might be included in special care management programs and the quality of care provided to him would be measured and tracked. Without diabetes on his problem list, he might receive none of these benefits.

In this study, the investigators developed an clinical decision support intervention that will identify patients with problem lists gaps. The investigators will alert providers of these likely gaps and offer providers the opportunity to correct them.

ELIGIBILITY:
Inclusion Criteria:

* Independent healthcare provider (physician, NP, PA)
* Practices at participating site

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptance | 6 months (May 2010-Nov2010)
  Of those providers who were shown (or who would have been shown, for the control group) the intervention, the number that added a problem across control and intervention groups.

SECONDARY OUTCOMES:
Problem list prevalence | pre and post intervention
  Number of patients with selected problems on their problem list pre and post intervention across intervention and control groups.
Problem list incidence | pre and post intervention
  For the conditions of interest, the percent of patients that had the problem added during the study period
Quality improvement based on problem list accuracy/completion | post intervention
  For those with problems added due to the intervention, the number of new triggered reminders or other clinical actions.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wright, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wright A, Pang J, Feblowitz JC, Maloney FL, Wilcox AR, McLoughlin KS, Ramelson H, Schneider L, Bates DW. Improving completeness of electronic problem lists through clinical decision support: a randomized, controlled trial. J Am Med Inform Assoc. 2012 Jul-Aug;19(4):555-61. doi: 10.1136/amiajnl-2011-000521. Epub 2012 Jan 3. PMID 22215056